CLINICAL TRIAL: NCT02251717
Title: A Phase 2, Open Label Study to Evaluate The Safety and Efficacy of Ledipasvir/Sofosbuvir (LDV/SOF) Fixed Dose Combination (FDC) Tablet for 12 or 24 Weeks in Kidney Transplant Recipients With Chronic HCV Infection
Brief Title: Safety and Efficacy of Ledipasvir/Sofosbuvir (LDV/SOF) Fixed Dose Combination (FDC) for 12 or 24 Weeks in Kidney Transplant Recipients With Chronic HCV Infection
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Gilead Sciences (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GS-US-337-1406; 2014-002121-35 (EudraCT Number)
Record Dates: First submitted 2014-09-25; First posted 2014-09-29 (Estimated); Results first posted 2017-11-17 (Actual); Last update posted 2018-11-19 (Actual); Status verified 2017-11

CONDITIONS: Hepatitis C Virus Infection
Keywords: renal transplant
MeSH Terms: conditions — Hepatitis C | interventions — ledipasvir, sofosbuvir drug combination

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- LDV/SOF 12 wk (Experimental): Participants will receive LDV/SOF FDC for 12 weeks.
  Interventions: Drug: LDV/SOF
- LDV/SOF 24 wk (Experimental): Participants will receive LDV/SOF FDC for 24 weeks.
  Interventions: Drug: LDV/SOF

INTERVENTIONS:
Drug: LDV/SOF — 90/400 mg FDC tablet administered orally once daily
  Other Names: Harvoni®; GS-5885/GS-7977

SUMMARY:
This study will evaluate the safety, tolerability, and antiviral efficacy of ledipasvir/sofosbuvir (LDV/SOF) fixed-dose combination (FDC) for 12 or 24 weeks in adults with chronic genotype 1 or genotype 4 hepatitis C virus (HCV) infection who have had a kidney transplant.

ELIGIBILITY:
Key Inclusion Criteria:

* Genotype 1 or 4 chronic HCV infection
* Have received a kidney transplant more than 6 months before the Baseline visit
* Cirrhosis determination
* Screening laboratory parameters within defined thresholds
* Use of two effective contraception methods if female of childbearing potential or sexually active male

Key Exclusion Criteria:

* Pregnant or nursing female or male with pregnant female partner
* Hepatocellular carcinoma (HCC) or other malignancy (with exception of certain -resolved skin cancers)
* History of clinically significant illness or any other medical disorder that may interfere with subject treatment, assessment or compliance with the protocol
* Planned or anticipated second kidney transplant

Note: Other protocol defined Inclusion/Exclusion criteria may apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 114 (Actual)
Dates: Start 2014-10-14 (Actual); Primary Completion 2016-03-24 (Actual); Study Completion 2016-06-16 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gilead Study Director, Study Director — Gilead Sciences
Locations (5):
- Vienna, Austria
- France (2):
  - Marseille
  - Paris
- Hanover, Germany
- Milan, Italy

IPD SHARING:
Plan to Share IPD: Yes
Qualified external researchers may request IPD for this study after study completion. For more information, please visit our website at http://www.gilead.com/research/disclosure-and-transparency.
Supporting Information: Study Protocol, SAP
Time Frame: 18 months after study completion
Access Criteria: A secured external environment with username, password, and RSA code.
URL: http://www.gilead.com/research/disclosure-and-transparency

REFERENCES:
- [Result] Colombo M, Aghemo A, Liu H, Dvory-Sobol H, Hyland RH, Yun C, Brainard DM, McHutchison JG, Bourliere M, Peck-Radosavljevic M, Manns M, Pol S. Ledipasvir/Sofosbuvir (LDV/SOF) for 12 or 24 Weeks Is Safe and Effective in Kidney Transplant Recipients With Chronic Genotype 1 or 4 HCV Infection. Journal of Hepatology. 2016;64 pp S183-S212. (GS 13, oral presentation).
- [Result] Colombo M, Aghemo A, Liu H, Zhang J, Dvory-Sobol H, Hyland R, Yun C, Massetto B, Brainard DM, McHutchison JG, Bourliere M, Peck-Radosavljevic M, Manns M, Pol S. Treatment With Ledipasvir-Sofosbuvir for 12 or 24 Weeks in Kidney Transplant Recipients With Chronic Hepatitis C Virus Genotype 1 or 4 Infection: A Randomized Trial. Ann Intern Med. 2017 Jan 17;166(2):109-117. doi: 10.7326/M16-1205. Epub 2016 Nov 15. PMID 27842383

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled at study sites in Europe. The first participant was screened on 14 October 2014. The last study visit occurred on 16 June 2016.
Pre-assignment Details: 130 participants were screened.
Groups:
- LDV/SOF 12 Weeks: Ledipasvir/sofosbuvir (Harvoni®; LDV/SOF) (90/400 mg) for 12 weeks in participants with chronic genotype 1 or 4 HCV infection who have had a kidney transplant
- LDV/SOF 24 Weeks: LDV/SOF (90/400 mg) for 24 weeks in participants with chronic genotype 1 or 4 HCV infection who have had a kidney transplant
Period: Overall Study
Arm/Group | LDV/SOF 12 Weeks | LDV/SOF 24 Weeks
Started | 57 | 57
Completed | 56 | 56
Not Completed | 1 | 1
Not completed — Adverse Event | 0 | 1
Not completed — Withdrew Consent | 1 | 0

BASELINE CHARACTERISTICS:
Population: Safety Analysis Set: participants who received at least 1 dose of study drug
Groups:
- LDV/SOF 12 Weeks: LDV/SOF (90/400 mg) for 12 weeks in participants with chronic genotype 1 or 4 HCV infection who have had a kidney transplant
- Total: Total of all reporting groups
Arm/Group | LDV/SOF 12 Weeks | LDV/SOF 24 Weeks | Total
Number analyzed (Participants) | 57 | 57 | 114
Age, Continuous [Mean (Standard Deviation); unit: years] | 54 (8.3) | 53 (10.0) | 53 (9.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 24 | 24 | 48
  Male | 33 | 33 | 66
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 4 | 5
  Not Hispanic or Latino | 56 | 53 | 109
  Unknown or Not Reported | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Black or African American | 2 | 2 | 4
  White | 54 | 53 | 107
  Asian | 1 | 1 | 2
  Other | 0 | 1 | 1
Region of Enrollment [Number; unit: participants]
  Austria | 9 | 15 | 24
  Italy | 32 | 17 | 49
  France | 15 | 21 | 36
  Germany | 1 | 4 | 5
HCV genotype [Count of Participants; unit: Participants]
  Genotype 1 | 51 | 53 | 104
  Genotype 4 | 6 | 4 | 10
Cirrhosis Status [Count of Participants; unit: Participants]
  No | 49 | 48 | 97
  Yes | 8 | 9 | 17
IL28b Status [Count of Participants; unit: Participants] — The CC, CT, and TT alleles are different forms of the IL28b gene.
  Participants
    CC | 14 | 18 | 32
    CT | 34 | 34 | 68
    TT | 9 | 5 | 14
Years From Most Recent Kidney Transplant [Mean (Standard Deviation); unit: years] | 12.1 (9.51) | 14.4 (9.66) | 13.2 (9.61)
HCV RNA [Mean (Standard Deviation); unit: log10 IU/mL] | 6.3 (0.63) | 6.2 (0.53) | 6.3 (0.58)
HCV RNA Category [Count of Participants; unit: Participants]
  < 800,000 IU/mL | 11 | 16 | 27
  ≥ 800,000 IU/mL | 46 | 41 | 87
Prior HCV Treatment Status [Count of Participants; unit: Participants]
  Treatment-Naive | 40 | 39 | 79
  Treatment-Experienced | 17 | 18 | 35

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Sustained Virologic Response (SVR) 12 Weeks After Discontinuation of Therapy (SVR12)
Description: SVR12 was defined as HCV RNA < the lower limit of quantitation (LLOQ; ie, 15 IU/mL) at 12 weeks after stopping study treatment.
Time Frame: Posttreatment Week 12
Population: Full Analysis Set: participants who were randomized into the study and received at least 1 dose of study drug
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | LDV/SOF 12 Weeks | LDV/SOF 24 Weeks
Number analyzed (Participants) | 57 | 57
percentage of participants | 100.0 [93.7 to 100.0] | 100.0 [93.7 to 100.0]

2. Primary Outcome: Percentage of Participants Who Permanently Discontinued Any Study Drug Due to an Adverse Event
Time Frame: Up to 24 weeks
Population: Safety Analysis Set: participants who received at least 1 dose of study drug
Measure: Number; unit: percentage of participants
Arm/Group | LDV/SOF 12 Weeks | LDV/SOF 24 Weeks
Number analyzed (Participants) | 57 | 57
percentage of participants | 1.8 | 0

3. Secondary Outcome: Percentage of Participants With SVR at 4 and 24 Weeks After Discontinuation of Therapy (SVR4 and SVR24)
Description: SVR4 and SVR24 were defined as HCV RNA < LLOQ at 4 and 24 weeks after stopping study treatment, respectively.
Time Frame: Posttreatment Weeks 4 and 24
Population: Full Analysis Set: participants who were randomized into the study and received at least 1 dose of study drug
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | LDV/SOF 12 Weeks | LDV/SOF 24 Weeks
Number analyzed (Participants) | 57 | 57
percentage of participants
  SVR4 | 100.0 [93.7 to 100.0] | 100.0 [93.7 to 100.0]
  SVR24 | 100.0 [93.7 to 100.0] | 100.0 [93.7 to 100.0]

4. Secondary Outcome: Percentage of Participants With Virologic Failure
Description: Virologic failure was defined as:
  * On-treatment virologic failure:
    * Breakthrough (confirmed HCV RNA ≥ LLOQ after having previously had HCV RNA < LLOQ while on treatment), or
    * Rebound (confirmed > 1 log10 IU/mL increase in HCV RNA from nadir while on treatment), or
    * Non-response (HCV RNA persistently ≥ LLOQ through 8 weeks of treatment)
  * Virologic relapse:
    * Confirmed HCV RNA ≥ LLOQ during the posttreatment period having achieved HCV RNA < LLOQ at last on-treatment visit.
Time Frame: Up to Posttreatment Week 24
Population: Full Analysis Set: participants who were randomized into the study and received at least 1 dose of study drug
Measure: Number; unit: percentage of participants
Arm/Group | LDV/SOF 12 Weeks | LDV/SOF 24 Weeks
Number analyzed (Participants) | 57 | 57
percentage of participants | 0 | 0

ADVERSE EVENTS:
Time Frame: Up to 24 weeks plus 30 days
Description: Safety Analysis Set: participants who received at least 1 dose of study drug
Arm/Group | LDV/SOF 12 Weeks | LDV/SOF 24 Weeks
All-Cause Mortality (participants affected / at risk) | 0/57 | 0/57
Serious Adverse Events (participants affected / at risk) | 5/57 | 8/57
Other Adverse Events (participants affected / at risk) | 23/57 | 36/57
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | LDV/SOF 12 Weeks (N=57) | LDV/SOF 24 Weeks (N=57)
Diarrhoea haemorrhagic (Gastrointestinal disorders) | 0 | 1
Erysipelas (Infections and infestations) | 1 | 0
Gastroenteritis (Infections and infestations) | 1 | 0
Urinary tract infection (Infections and infestations) | 0 | 1
Incisional hernia (Injury, poisoning and procedural complications) | 0 | 1
Shunt thrombosis (Injury, poisoning and procedural complications) | 0 | 1
Blood creatinine increased (Investigations) | 0 | 1
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 0 | 1
Papillary thyroid cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Syncope (Nervous system disorders) | 1 | 0
Suicide attempt (Psychiatric disorders) | 1 | 0
Acute kidney injury (Renal and urinary disorders) | 1 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Arteriovenous shunt operation (Surgical and medical procedures) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | LDV/SOF 12 Weeks (N=57) | LDV/SOF 24 Weeks (N=57)
Anaemia (Blood and lymphatic system disorders) | 1 | 3
Abdominal pain (Gastrointestinal disorders) | 0 | 4
Diarrhoea (Gastrointestinal disorders) | 3 | 5
Nausea (Gastrointestinal disorders) | 3 | 3
Vomiting (Gastrointestinal disorders) | 3 | 1
Asthenia (General disorders) | 8 | 8
Fatigue (General disorders) | 4 | 7
Oedema peripheral (General disorders) | 0 | 3
Bronchitis (Infections and infestations) | 0 | 3
Nasopharyngitis (Infections and infestations) | 0 | 5
Urinary tract infection (Infections and infestations) | 4 | 4
Hyperuricaemia (Metabolism and nutrition disorders) | 2 | 5
Arthralgia (Musculoskeletal and connective tissue disorders) | 4 | 0
Headache (Nervous system disorders) | 9 | 13
Somnolence (Nervous system disorders) | 1 | 3
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 3
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 4
Haematoma (Vascular disorders) | 0 | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
After conclusion of the study and without prior written approval from Gilead, investigators in this study may communicate, orally present, or publish in scientific journals or other media only after the following conditions have been met:

* The results of the study in their entirety have been publicly disclosed by or with the consent of Gilead in an abstract, manuscript, or presentation form; or
* The study has been completed at all study sites for at least 2 years